CLINICAL TRIAL: NCT04433286
Title: COVID-19 - Implications on Surgeons' Burnout and Career Satisfaction
Acronym: SURG-SAT-19
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mostafa shalaby, MD, MSc, PhD, Dr, Mansoura University
Other Study IDs: SURG RES COL 1
Record Dates: First submitted 2020-06-10; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Physical Stress; Career Burnout; Satisfaction
MeSH Terms: conditions — Burnout, Professional; Personal Satisfaction | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — This is a cross-sectional survey which will be distributed online between surgeons. The survey was proposed by a consensus of consultants of surgery and revised by an improvement consultant. It consists of a semi-structured questionnaire that is provided in English language. A subsequent translation in different Language will provided based on geographical distribution. The survey will be conducted online through an online survey development cloud-based software (SurveyMonkey®; San Mateo, CA, USA). Participants will be aware of the nature of the survey and informed that they will be listed as co-authors. Collected data will be confidential and anonymous.
  The first sector of the questionnaire includes trainee demographics and baseline characteristics. Then the questionnaire aims to compare the trainee experience before and after the pandemic with focus on research activities, clinical, and surgical practice.

SUMMARY:
This is a cross-sectional survey which will be distributed online between surgeons. The survey was proposed by a consensus of consultants of surgery and revised by an improvement consultant. It consists of a semi-structured questionnaire that is provided in English language. The survey will be conducted online through an online survey development cloud-based software (SurveyMonkey®; San Mateo, CA, USA). Participants will be aware of the nature of the survey and informed that they will be listed as co-authors. Collected data will be confidential and anonymous.

The first sector of the questionnaire includes trainee demographics and baseline characteristics. Then the questionnaire aims to compare the trainee experience before and after the pandemic with focus on research activities, clinical, and surgical practice.

DETAILED DESCRIPTION:
This is a cross-sectional survey which will be distributed online between surgeons. The survey was proposed by a consensus of consultants of surgery and revised by an improvement consultant. It consists of a semi-structured questionnaire that is provided in English language. A subsequent translation in different Language will provided based on geographical distribution. The survey will be conducted online through an online survey development cloud-based software (SurveyMonkey®; San Mateo, CA, USA). Participants will be aware of the nature of the survey and informed that they will be listed as co-authors. Collected data will be confidential and anonymous.

The first sector of the questionnaire includes trainee demographics and baseline characteristics. Then the questionnaire aims to compare the trainee experience before and after the pandemic with focus on research activities, clinical, and surgical practice.

Statistical analyses will be performed using SPSS v. 20. Data distribution will be tested for normality using the Kolmogorov-Smirnov test and the Shapiro-Wilk test. Categorical variables will be expressed as group percentages and will be compared for independent samples using the Chi-square test. Continuous data of the survey will be presented as medians with ranges or means and standard deviations. A comparison of continuous data will be compared for independent samples using the T-test or Mann-Whitney test according to the data distribution. Spearman correlation coefficient will be used for further assessment of the strength of the association between variables. The statistical significance level will be set at <0.05.

ELIGIBILITY:
Inclusion Criteria:

* The Survey is targeting surgeons of all specialities; Cardiothoracic, General, Neurosurgery, Oral and Maxillofacial, Otolaryngology, Pediatric, Plastic, Trauma and Orthopedic, Urology, and Vascular Surgery. Furthermore, Gynecological Oncology and Urogynecology surgeons are invited.

Exclusion Criteria:

* other specialities other than surgery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Surgeons of all specialities; Cardiothoracic, General, Neurosurgery, Oral and Maxillofacial, Otolaryngology, Pediatric, Plastic, Trauma and Orthopedic, Urology, and Vascular Surgery. Furthermore, Gynecological Oncology and Urogynecology surgeons are invited.
  Both sex.
  All over the globe.
  Any level of experiences.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-06-15 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Burnout before COVID-19 and during COVID-19 | 1 year before COVID-19 versus during the COVID-19 pandemic (Mrach-June 2020)
  A questionnaire designed based on the literature review to assess Burnout
Change in Job satisfaction before COVID-19 and during COVID-19 | 1 year before COVID-19 versus during the COVID-19 pandemic (Mrach-June 2020)
  A questionnaire designed based on the literature review to assess Job satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Shalaby, MD, MSc, PhD, Principal Investigator — Mansoura Faculty of Medicine; Hosam Hamed, MD, MSc, PhD, Study Chair — Mansoura Faculty of Medicine; Ahmed M Elsheikh, MD,MBA,CMQOE, Study Director — Security Forces Program Hospital
Locations (1):
- Faculty of Medicine Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shalaby M, ElSheikh AM, Hamed H; SURG-SAT-19 Collaborative Group. Burnout among surgeons before and during the SARS-CoV-2 pandemic: an international survey. BMC Psychol. 2024 Jan 25;12(1):48. doi: 10.1186/s40359-023-01517-4. PMID 38273390